CLINICAL TRIAL: NCT03957330
Title: Therapeutics Moderators of Therapist-assisted Internet-delivered Cognitive Behavior Therapy for Depression and Anxiety
Brief Title: Therapeutic Moderators of Therapist-assisted Internet-delivered Cognitive Behavior Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-038
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Internet-delivered cognitive behaviour therapy; Randomized controlled trial; Therapist contact; Online therapy; Community mental health
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are told about the nature of their treatment but not about the exact nature of all the conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Community Mental Health Clinic (Experimental): In this arm, clients will be assigned to therapists working in a community mental health clinic in Saskatchewan where the focus of the setting is primarily on face-to-face treatment and ICBT makes up a small component of the workload in the clinic.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- Once a week therapist contact (Experimental): In once a week treatment, therapists will email their clients once a week on a pre-determined day.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- Reflection Questionnaire (Experimental): In the reflection questionnaire, patients will be asked to complete the following questions five times during the treatment period (beginning lesson 2-5 and then at the point they complete post-questionnaires):
  1. How much of the lesson were you able to review?
  2. How much effort were you able to put into the lesson?
  3. How difficult was the lesson?
  4. Please share any difficulties you had with the lesson.
  5. How understandable was the lesson?
  6. How helpful did you find the lesson?
  7. Please describe an example of what you learned.
  8. To what extent have you continued to use strategies from previous lessons
  9. If applicable, please provide an example of what you are working on from previous lessons
  10. Please indicate which Additional Resources you reviewed this week.
  11. If applicable, please share any skills you are working on from the Additional Resources.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- Specialized Internet Therapy Clinic (Experimental): In this arm, clients will be assigned to therapists working in a specialized internet therapy clinic where the therapists only deliver ICBT.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- Twice a week therapist contact (Experimental): In twice a week treatment, therapists will email their clients twice a week on pre-determined days.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- No Reflection Questionnaire (Experimental): In this arm, no reflection questions will be asked of clients receiving ICBT.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behaviour therapy — All clients will receive the Wellbeing Course developed at Macquarie University, Australia. The Wellbeing Course is a transdiagnostic Internet-delivered cognitive behaviour intervention targeting symptoms of depressive and anxiety disorders. It comprises 5 online lessons targeting: 1) symptom identification and the cognitive behavioural model; 2) thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling; 4) graduated exposure; and 5) relapse prevention. Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills) and include homework activities. Lessons are released gradually in a standardized order over 8 weeks. Phone calls will only be made if there is a significant clinical issue requiring therapist attention that cannot be addressed over email (e.g., sudden increase in symptoms). Therapists will spend ~15 mins. per week/per client.

SUMMARY:
Depression and anxiety are common and prevalent conditions that often go untreated. In an attempt to increase timely and accessible psychological treatment, Internet-delivered cognitive behavioural therapy (ICBT) has emerged. ICBT involves delivering therapeutic content via structured online lessons. This is often combined with therapist guidance, such as once per week contact via secure messaging or phone calls over several months. Over the past several years, the investigators have been studying the efficacy of ICBT for symptoms of depression and anxiety and found ~70% of patient's fully complete treatment and demonstrate large improvement in symptoms. Although outcomes of ICBT are very impressive, there is some room for improvement in terms of completion rates and outcomes.

In this three-factorial randomized controlled trial, the investigators aim to contribute to the literature by examining whether the efficacy of ICBT in routine practice is moderated by amount of contact (once versus twice a week), inclusion of homework reflection questionnaire (yes vs no) and location of therapist (specialized unit vs community mental health clinic). Follow-up measures will be carried out at 3, 6 and 12 months after randomization. Primary outcomes are reduced anxiety and depression. Secondary outcomes include psychological distress, panic, social anxiety, trauma, health anxiety, quality of life, disability, intervention usage (e.g., completion rates, log-ins, emails sent), satisfaction, therapeutic alliance, and costs (e.g., health care utilization).

DETAILED DESCRIPTION:
Based on past research of ICBT in routine care, patients and therapists have expressed an interest in "personalizing" the delivery of ICBT, for example, by increasing the amount of therapist support available (from once a week to twice a week) to reflect the unique needs and preferences of the patients. Patients also express an interest in personalizing "therapy messages". One current barrier to offering more personalized messages, however, is that patients do not consistently provide information on their use of new treatment strategies, as well as strengths and challenges of using strategies. As a result, therapists find it difficult to personalize their messages. One method of overcoming this difficulty is to systematically ask patients to reflect on their use of treatment strategies (e.g., monitoring thoughts, challenging thoughts, controlled breathing, pleasant activities, and exposure) through questionnaires rather than relying on patients to provide this information in emails. Another factor that could moderate ICBT efficacy is therapist location. Some therapists who provide ICBT work in a specialized unit where there is primary focus on ICBT and daily attention to following ICBT guidelines. Other therapists deliver ICBT from community mental health clinics where the primary focus of the setting is on face-to-face care and there is lower familiarity with ICBT. It is possible that ICBT may be more effectively delivered in a setting where the primary focus is on ICBT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Endorse symptoms of anxiety or depression
* Resident of Saskatchewan
* Access to a computer and the Internet

Exclusion Criteria:

* Have a severe psychiatric illness (e.g. psychosis)
* Assessed as being at high risk of suicide
* Report severe problems with alcohol or drugs
* Report severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) | Baseline, weeks 2, 4, 5, 7, 8 and 3-, 6-, and 12-month follow-up
  Change in depression symptoms. 9 items are summed into a total score, with scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline, weeks 2, 4, 5, 7, 8, and 3-, 6-, and 12-month follow-up
  Change in anxiety symptoms. 7 items are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.

SECONDARY OUTCOMES:
Panic Disorder Severity Scale Self-report | Time Frame: Baseline, week 8, and 3-, 6-, and 12-month follow-up
  Change in panic symptoms. Items are summed into a total score. Total scores range between 0 and 28, with higher scores representing more severe self-reported symptoms of panic.
Social Interaction Anxiety Scale (6 items) and Social Phobia Scale-Short form (6 items) | Time Frame: Baseline, Week 8, 3-, 6-, and 12-month follow-up
  Change in social anxiety symptoms. Items from the two measures are summed into a total score. Total scores range between 0 and 48, with higher scores representing more severe self-reported symptoms of social anxiety
PTSD Check List 5 | Baseline, week 8 and 3-, 6-, and 12-month follow-up
  Change in post-traumatic symptoms. The measure consists of 20 questions rated 0 to 4; higher scores indicate more trauma symptoms The first section assesses for exposure to a traumatic event using a checklist question. If the client endorses exposure to a traumatic event, they are provided the second section, which assesses severity of trauma symptoms. Items are summed into a total score, which can range between 0 and 80. Higher scores represent more severe self-reported symptoms of trauma.
Short Health Anxiety Inventory-14 | Baseline, week 8 and 3-, 6-, and 12-month follow-up
  Change in health anxiety. 14 items with higher scores indicating higher levels of self-reported health anxiety.
Kessler Psychological Distress | Baseline, week 8, and 3-, 6-, and 12-month follow-up
  Change in psychological distress. Measured by 10-item scale rated 0 to 4; total score is created by summing items; higher scores signify greater psychological distress
Quality of life questionnaire (EQ-ED-5L) | Baseline, week 8, and 3-, 6-, and 12-month follow-up
  Change in quality of life. Items are summed into six sub-total scores. The first five sub-total scores respectively assess various domains of quality of life (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).
  Each of the five sub-total scores range between 1 and 5, with higher scores representing greater self-reported severity and impairment in these various domains. The last sub-total score provides an overall index of health and can range between 0 and 100, with higher scores representing better self-reported health.
Sheehan Disability Scale 3-item | Baseline, week 8, and 3-, 6-, and 12-month follow-up
  Change in disability. Measure consists of 3 items rated 0 to 10 and summed to create total score, with higher scores indicating greater disability
Treatment Inventory of Costs in Psychiatric Patients (TIC-P) Adapted for Canada | Baseline and 3-, 6-, and 12-month follow-up
  Change in treatment costs. A series of yes and no, rating, and frequency questions that are designed to ascertain the volume of medical consumption and productivity losses associated with mental health problems. Questions are independently analyzed and, therefore, the TIP-C does not include a total score.
Treatment Credibility Questionnaire | Baseline, week 8, and 3-month follow-up
  Change in treatment credibility. 4 items are summed into a total score. Higher scores representing greater perceptions of ICBT credibility.
Working Alliance Inventory Short-Form | Baseline, week 8, and 3-, 6-, and 12-month follow-up
  Measures therapeutic alliance. Scores are summed into three sub-total scores, which respectively assess various domains of the therapeutic relationship (i.e., goal, task, and bond). Sub-total scores each range between 5 and 20, with higher scores representing better therapeutic relationship in each of the three domains assessed.
Treatment Engagement | Week 8
  Measured by: number of lessons completed, number of days of access, number of emails sent to therapist, number of phone calls with therapist, number of emails from therapist to client, total words emailed to therapist, total words emailed from therapist to patient
Treatment Satisfaction and Negative Effects Questionnaires | Week 8
  Measure includes 19 questions assessing satisfaction with various aspects of Internet-CBT and also negative effects of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

REFERENCES:
- [Derived] Sapkota RP, Peynenburg V, Dear BF, Titov N, Hadjistavropoulos HD. Engagement with homework in an Internet-delivered therapy predicts reduced anxiety and depression symptoms: A latent growth curve analysis. J Consult Clin Psychol. 2023 Feb;91(2):112-117. doi: 10.1037/ccp0000775. Epub 2022 Nov 17. PMID 36395032